CLINICAL TRIAL: NCT01782872
Title: Analgesia After Total Shoulder Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-014
Record Dates: First submitted 2012-09-24; First posted 2013-02-04 (Estimated); Results first posted 2016-05-18 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-04

CONDITIONS: Total Shoulder Arthroplasty
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Interscalene Block (ISB) - 0.375% Ropivacaine + additives (Active Comparator)
  Interventions: Procedure: Interscalene Block (ISB) - 0.375% Ropivacaine + additives
- Interscalene Block (ISB) - 0.2% Ropivacaine + additives (Active Comparator)
  Interventions: Procedure: Interscalene Block (ISB) - 0.2% Ropivacaine + additives
- Interscalene Block (ISB) - 0.1% Ropivacaine + additives (Active Comparator)
  Interventions: Procedure: Interscalene Block (ISB) - 0.1% Ropivacaine + additives
- Interscalene Block (ISB) - Systemic Control (Active Comparator)
  Interventions: Procedure: Interscalene Block (ISB) - Systemic Control

INTERVENTIONS:
Procedure: Interscalene Block (ISB) - 0.375% Ropivacaine + additives — Ultrasound-guided single-injection ISB: ropivacaine 0.375% + (clonidine [100 mcg] + dexamethasone [4 mg] + buprenorphine [150 mcg]); Intravenous (IV): saline
  Arms: Interscalene Block (ISB) - 0.375% Ropivacaine + additives
Procedure: Interscalene Block (ISB) - 0.2% Ropivacaine + additives — Ultrasound-guided single-injection ISB: ropivacaine 0.2% + (clonidine [100 mcg] + dexamethasone [4 mg] + buprenorphine [150 mcg]); Intravenous: saline
  Arms: Interscalene Block (ISB) - 0.2% Ropivacaine + additives
Procedure: Interscalene Block (ISB) - 0.1% Ropivacaine + additives — Ultrasound-guided single-injection ISB: ropivacaine 0.1% + (clonidine [100 mcg] + dexamethasone [4 mg] + buprenorphine [150 mcg]); Intravenous: saline
  Arms: Interscalene Block (ISB) - 0.1% Ropivacaine + additives
Procedure: Interscalene Block (ISB) - Systemic Control — Ultrasound-guided single-injection ISB: ropivacaine 0.375%; Intravenous: clonidine (100 mcg) + dexamethasone (4 mg) + buprenorphine (150 mcg)
  Arms: Interscalene Block (ISB) - Systemic Control

SUMMARY:
The purpose of this study is to determine which medication(s) should be included in the interscalene nerve block (an injection of local anesthetic [numbing medicine] near nerves in the shoulder) for patients undergoing total shoulder arthroplasty (shoulder replacement). The ideal nerve block would reduce pain after shoulder surgery without causing a great deal of muscle weakness.

DETAILED DESCRIPTION:
All patients will receive an intravenous pain pump (patient-controlled analgesia) and a nerve block with long-lasting local anesthetic. The three study groups will receive additives (clonidine, dexamethasone, buprenorphine plus local anesthetic) in the nerve block that may reduce postoperative pain. One of the study groups uses the usual concentration of local anesthetic, while the other two study groups use reduced concentrations of local anesthetic. Follow-up with study patients begins on the day of surgery and continues through postoperative day 2. Seen twice daily, patients will be asked about their pain and assessed for sensory function and strength of their shoulder muscle and hand grip.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis
* Primary total shoulder arthroplasty
* Age 18 to 80 years old
* Planned use of general anesthesia
* Planned use of a brachial plexus nerve block for postoperative analgesia
* Ability to follow study protocol

Exclusion Criteria:

* Patients younger than 18 years old and older than 80
* Allergy or intolerance to one of the study medications
* Patients with an American Society of Anesthesiologists (ASA) physical status of IV
* Patients with insulin-dependent diabetes
* Patients with hepatic (liver) failure
* Patients with chronic renal (kidney) failure
* Bradycardia (heart rate < 50) or hypotension (systolic blood pressure < 90 mmHg)
* Chronic opioid use (taking opioids for longer than 3 months) (or active diagnosis of complex regional pain syndrome [CRPS]/reflex sympathetic dystrophy [RSD])
* Lack of English fluency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques T YaDeau, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- High Dose: Interscalene Block (ISB) - 0.375% Ropivacaine + additives: Ultrasound-guided single-injection ISB: ropivacaine 0.375% + (clonidine [100 mcg] + dexamethasone [4 mg] + buprenorphine [150 mcg]); Intravenous (IV): saline
- Medium Dose: Interscalene Block (ISB) - 0.2% Ropivacaine + additives: Ultrasound-guided single-injection ISB: ropivacaine 0.2% + (clonidine [100 mcg] + dexamethasone [4 mg] + buprenorphine [150 mcg]); Intravenous: saline
- Low Dose: Interscalene Block (ISB) - 0.1% Ropivacaine + additives: Ultrasound-guided single-injection ISB: ropivacaine 0.1% + (clonidine [100 mcg] + dexamethasone [4 mg] + buprenorphine [150 mcg]); Intravenous: saline
- Control: Interscalene Block (ISB) - Systemic Control: Ultrasound-guided single-injection ISB: ropivacaine 0.375%; Intravenous: clonidine (100 mcg) + dexamethasone (4 mg) + buprenorphine (150 mcg)
Period: Overall Study
Arm/Group | High Dose | Medium Dose | Low Dose | Control
Started | 20 | 20 | 20 | 20
Completed | 20 | 19 | 20 | 19
Not Completed | 0 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose | Medium Dose | Low Dose | Control | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8) | 64 (9) | 69 (7) | 68 (7) | 67 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 15 | 10 | 47
  Male | 7 | 11 | 5 | 10 | 33
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 20 | 20 | 80
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28 (4) | 25 (3) | 27 (4) | 31 (6) | 28 (5)

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale (NRS) Pain Score With Movement
Description: Pain with movement at 24 hours from the nerve block (scale of 0-10; 0 = no pain, 10 = worst possible pain)
Time Frame: 24 hours after the interscalene block is given
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Dose | Medium Dose | Low Dose | Control
Number analyzed (Participants) | 20 | 19 | 20 | 19
units on a scale | 4.5 (3.0) | 3.4 (1.8) | 4.2 (2.4) | 4.9 (2.5)

2. Secondary Outcome: Duration of Analgesia From Interscalene Nerve Block
Description: Median time until a patient needed to take opioid pain medication
Time Frame: Postoperative day 1 at 8AM & 5PM, postoperative day 2 at 8AM & 5PM
Population: Patients who were able to provide actual or estimates of time until they first needed to use pain medication were included in this analysis.
Measure: Mean (Standard Error); unit: hours
Arm/Group | High Dose | Medium Dose | Low Dose | Control
Number analyzed (Participants) | 16 | 17 | 17 | 20
hours | 21.3 (1.0) | 16.8 (1.6) | 18.2 (1.9) | 16.4 (1.4)

3. Secondary Outcome: Numeric Rating Scale (NRS) Pain Scores at Rest
Description: Assessment of NRS pain scores (scale of 0-10; 0 = no pain, 10 = worst possible pain) at rest
Time Frame: Preop
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | High Dose | Medium Dose | Low Dose | Control
Number analyzed (Participants) | 20 | 19 | 20 | 19
units on a scale | 3.0 [1.7 to 5.5] | 3.2 [1.9 to 6.0] | 3.0 [1.0 to 4.6] | 4.9 [2.9 to 6.7]

4. Secondary Outcome: Middle Deltoid
Description: A physical assessment will be done to determine the strength of the middle deltoid muscle in the operative arm using a dynamometer
Time Frame: 24 hours after surgery
Population: Patients who agreed to the measurements were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: kgf
Arm/Group | High Dose | Medium Dose | Low Dose | Control
Number analyzed (Participants) | 18 | 17 | 18 | 19
kgf | 2.8 [1.7 to 4.2] | 1.5 [1.3 to 2.2] | 2.2 [2.0 to 3.2] | 1.8 [1.4 to 2.2]

ADVERSE EVENTS:
Arm/Group | High Dose | Medium Dose | Low Dose | Control
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes